CLINICAL TRIAL: NCT01836666
Title: Effects on Health Related Quality of Life Among Patients With Chronic Pain by Interventional Pain Management
Status: Completed | Type: Observational
Sponsor: Eques Indolor AB (Other)
Responsible Party: Sponsor
Other Study IDs: SE-Dnr-2012-446-31M-1
Record Dates: First submitted 2013-04-16; First posted 2013-04-22 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
How are the health related quality of life among patients with chronic pain effected by interventional pain managment?

Hypothesis:

Health related quality of life can be improved by interventional pain management both among patients with localizable pain focuses and among patients among whom no pain focuses can be found.

Method:

Health related quality of life using EQ-5D and EQ-VAS is registered at first visit, at the time of treatment for pain focuses an during the following 12 months.

ELIGIBILITY:
Inclusion Criteria:

All patients

Exclusion Criteria:

-

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to a specialized interventional pain management clinic in northen sweden
Sampling Method: Non-Probability Sample
Enrollment: 873 (Actual)
Dates: Start 2008-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
EQ-VAS | 1 year
  EQ-VAS is measured at first visit, at time for treatment and 3, 6 and 12 months after treatment. EQ-VAS gives a value of quality of life, and mainly used to verify the results achieved from EQ-5D since it is not possible to calculate QALY from EQ-VAS
EQ-5D | 1 year
  EQ-5D is assessed at first visit, at time for treatment and 3, 6 and 12 months after treatment. Quality of life is calculated from EQ-5D using the TTO-valuated UK value sets. This value can also be used for calculation of QALY, Quality adjusted life years.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hambraeus, MD, Principal Investigator
Locations (1):
- Smärtkliniken Eques Indolor, Vallentuna, Sweden